CLINICAL TRIAL: NCT06675136
Title: Phase 1 Trial of Nab-Paclitaxel PIPAC (Pressurized Intraperitoneal Aerosolized Chemotherapy) Given in Combination With Second-Line Therapy for Gastric Cancer With Peritoneal Metastases
Brief Title: Nab-Paclitaxel PIPAC in Combination With Paclitaxel and Ramucirumab for the Treatment of Stomach Cancer With Peritoneal Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24445; NCI-2024-08883 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24445 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Clinical Stage IVB Gastric Cancer AJCC v8; Metastatic Gastric Adenocarcinoma; Metastatic Malignant Neoplasm in the Peritoneum
MeSH Terms: interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Paclitaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nab-paclitaxel PIPAC, paclitaxel, ramucirumab) (Experimental): Patients receive nab-paclitaxel PIPAC IP over 40 minutes on day 1 and SOC paclitaxel IV over 60 minutes on days 15, 22, 29, 43, and 50 and ramucirumab IV over 30-60 minutes on days 15, 29 and 43 of each cycle. Cycles repeat every 8 weeks (56 days) for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may then continue SOC paclitaxel IV on days 1, 8, and 15 and ramucirumab IV on days 1 and 15 of each cycle per physician as deemed appropriate. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, tumor biopsy, and CT or MRI throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Medical Device Usage and Evaluation; Drug: Nab-paclitaxel; Drug: Paclitaxel; Other: Questionnaire Administration; Biological: Ramucirumab

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Medical Device Usage and Evaluation — Given PIPAC
Drug: Nab-paclitaxel — Given IP
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Questionnaire Administration — Ancillary studies
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC 1121B; IMC-1121B; IMC1121B; LY 3009806; LY-3009806; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase I trial tests the safety, side effects and best dose of nab-paclitaxel pressurized intraperitoneal aerosolized chemotherapy (PIPAC) in combination with second-line chemotherapy, paclitaxel and ramucirumab, and tests how well they work in treating stomach cancer that has spread from where it first started to the tissue that lines the abdominal wall and organs (peritoneal metastases). Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Nab-paclitaxel is an albumin-stabilized nanoparticle formulation of paclitaxel which may have fewer side effects and work better than other forms of paclitaxel. PIPAC delivers chemotherapy, such as nab-paclitaxel, that has been turned into a fine mist (aerosolized) at a high pressure directly into the abdominal cavity. Aerosolized chemotherapy delivered directly into the peritoneal space has been shown to deliver higher drug concentrations to the tumor. Ramucirumab is a monoclonal antibody that may prevent the growth of new blood vessels that tumors need to grow. Giving nab-paclitaxel PIPAC in combination with paclitaxel and ramucirumab may be safe, tolerable, and/or effective in treating gastric cancer patients with peritoneal metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of nab-paclitaxel PIPAC when given in combination with standard-of-care second-line systemic therapy (paclitaxel, ramucirumab).

II. To assess the safety and tolerability of nab-paclitaxel PIPAC plus systemic paclitaxel and ramucirumab, and accompanying dose modification plan, by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. To evaluate the anti-tumor activity of nab-paclitaxel when given in combination with standard-of-care second-line systemic therapy (paclitaxel, ramucirumab), as assessed by:

Ia. Response Evaluation Criteria in Solid Tumors (RECIST), if available, version 1.1 via computed tomography (CT) scan at baseline and every 8 weeks until disease progression; Ib. Peritoneal Regression Grading Score (PRGS) via biopsy at each PIPAC cycle (both pre-PIPAC and post-PIPAC peritoneal samples will be obtained); Ic. Peritoneal Carcinomatosis Index (PCI) at the time of laparoscopy; and Id. Overall survival (OS) and progression-free survival (PFS) estimates at 6-months, 1-year and 2-years.

II. To estimate the PIPAC technical failure rate. III. To characterize and evaluate peritoneal tumor associated complications. IV. To characterize and evaluate post-operative surgical complications by Clavien-Dindo classification evaluated at 30 days after each PIPAC technical failure rate.

V. To evaluate patient-reported health state/quality of life and symptoms before treatment and at 6, 12, 18, and 24 weeks/off study, as measured by the European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) and MD Anderson Symptom Inventory (MDASI).

EXPLORATORY OBJECTIVES:

I. Characterize the peritoneal tumor and immune tumor microenvironment changes in response to therapy.

II. Evaluate the pharmacokinetics of nab-paclitaxel PIPAC. III. Evaluate patients' quality of life during nab-paclitaxel PIPAC plus systemic therapy.

OUTLINE: This is a dose-escalation study of nab-paclitaxel PIPAC in combination with paclitaxel and ramucirumab followed by a dose-expansion study.

Patients receive nab-paclitaxel PIPAC intraperitoneally (IP) over 40 minutes on day 1 and standard of care (SOC) paclitaxel intravenously (IV) over 60 minutes on days 15, 22, 29, 43, and 50 and ramucirumab IV over 30-60 minutes on days 15, 29 and 43 of each cycle. Cycles repeat every 8 weeks (56 days) for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may then continue SOC paclitaxel IV on days 1, 8, and 15 and ramucirumab IV on days 1 and 15 of each cycle per physician as deemed appropriate. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection, tumor biopsy, and CT or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 4 weeks, then every 3 months for year 1 followed by every 6 months until progression or initiation of a new systemic anti-cancer therapy or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have failed first-line systemic therapy (fluorouracil, leucovorin calcium, oxaliplatin [FOLFOX] with or without immunotherapy, or other fluoropyrimidine and platinum-based therapy)

  * Prior immunotherapy allowed
  * Up to 4 cycles of second-line therapy allowed if no progression is documented
* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed gastric adenocarcinoma
* Visible peritoneal metastatic disease on cross-sectional imaging or diagnostic laparoscopy (does not have to be measurable by RECIST 1.1)
* Fully recovered from acute toxic effects (except alopecia, hearing loss, or non-clinically significant laboratory abnormalities) ≤ grade 1 of prior anti-cancer therapy
* The patient's urinary protein is ≤ 1+ on dipstick or routine urinalysis. If urine dipstick or routine analysis indicates proteinuria ≥ 2+, then a 24-hour urine must be collected and must demonstrate < 1000mg protein in 24 hours
* Complete medical history and physical exam (within 28 days prior to day 1 of protocol therapy)
* Absolute neutrophil count (ANC) ≥ 1,500/mcL (within 28 days prior to day 1 of protocol therapy)
* Platelets ≥ 100,000/mcL (within 28 days prior to day 1 of protocol therapy)
* Hemoglobin ≥ 8 g/dL (within 28 days prior to day 1 of protocol therapy)
* Serum albumin ≥ 2.8 g/dL (within 28 days prior to day 1 of protocol therapy)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease, then direct bilirubin < 1.5 mg/dL) (within 28 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) ≤ 5 x ULN (within 28 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) ≤ 5 x ULN (within 28 days prior to day 1 of protocol therapy)
* International normalized ratio (INR) ≤ 1.5 x ULN (within 28 days prior to day 1 of protocol therapy)
* Prothrombin time (PT) ≤ 1.5 x ULN (within 28 days prior to day 1 of protocol therapy)
* Partial thromboplastin time (PTT) ≤ 1.5 x ULN (within 28 days prior to day 1 of protocol therapy)
* Calculated creatinine clearance of ≥ 45 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 28 days prior to day 1 of protocol therapy)
* Seronegative for HIV antigen (Ag)/antibody (Ab) combo (within 28 days prior to day 1 of protocol therapy)

  * If seropositive, patient may be eligible if they are stable on antiretroviral therapy, have a CD4 T cell count ≥ 200/µL, and have an undetectable viral load
* Documented virology status of hepatitis, confirmed by hepatitis B virus (HBV) and hepatitis C virus (HCV) tests (within 28 days prior to day 1 of protocol therapy)

  * For patients with active HBV, HBV deoxyribonucleic acid (DNA) < 500 IU/mL during screening, initiation of anti-HBV treatment at least 14 days prior to day 1 of cycle 1, and willingness to continue anti-HBV treatment during the study (per standard of care)
  * If seropositive for HCV, nucleic acid quantification must be performed. Viral load must be undetectable
* WOMEN OF CHILDBEARING POTENTIAL (WOCBP): Negative urine or serum pregnancy test (within 28 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control (e.g., licensed hormonal/barrier methods or surgery intended to prevent pregnancy [or with a side effect of pregnancy prevention]) or abstain from heterosexual activity for the course of the study through at least 14 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Intolerance to taxanes
* Bowel obstruction requiring exclusive total parenteral nutrition
* Any history of, or current, brain or subdural metastases
* Life expectancy < 3 months
* Treatment with therapeutic oral or IV antibiotics within 14 days prior to day 1 cycle 1 of treatment

  * Patients receiving prophylactic antibiotics are eligible, provided the signs of active infection have resolved
* Any prior malignancy except adequately treated basal or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for two years
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents (taxanes, etc.)
* Clinically significant uncontrolled illness such as uncontrolled hypertension (HTN)
* History of arterial thromboembolic events such as myocardial infarction (MI), cerebrovascular accident (CVA)
* History of gastrointestinal (GI) perforation
* FEMALES ONLY: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2029-01-14 (Estimated); Study Completion 2029-01-14 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 6 weeks after the first pressurized intraperitoneal aerosolized chemotherapy (PIPAC) treatment
  Will be evaluated and graded based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Toxicities will be summarized by type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment, and reversibility or outcome. Rates and associated 95% Clopper and Pearson binomial confidence limits will be estimated.

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events (AEs) | Up to 4 weeks after last dose of nab-paclitaxel
  Will be evaluated and graded based on NCI CTCAE v 5.0. The number and percent of patients with AEs will be tabulated by system organ class and preferred term using the Medical Dictionary for Regulatory Activities preferred term dictionary. The tabulations will be generated so that the number and percent of patients with events in each severity, relatedness, and serious category can be obtained for each preferred term. Listings and narratives will be provided for deaths on study, serious AEs, DLTs, and events leading to discontinuation of treatment.
Incidence of post-operative surgical complications | At 4 weeks post-PIPAC procedure
  Will be evaluated using Clavien-Dindo classification. Results will be strictly descriptive in nature.
Objective response rate (ORR) | Up to 2 years
  Will be evaluated according to Response Evaluation Criteria in Solid Tumors v 1.1. ORR will be defined as the percentage of evaluable patients who have achieved complete response (CR), partial response (PR), or stable disease (SD). Rates and associated 95% Clopper and Pearson binomial confidence limits will be estimated.
Peritoneal Carcinomatosis Index (PCI) | At time of laparoscopy
  PCI will be defined as the percentage of evaluable patients who have achieved CR, PR, or SD. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson
Peritoneal Regression Grading Score (PRGS) | At baseline and post-PIPAC, assessed up to 2 years
  PRGS will be defined as the percentage of evaluable patients who have achieved a decrease in the PRGS over successive biopsies. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson
Progression-free survival (PFS) | From first PIPAC to progression of disease, assessed up to 2 years
  PFS will be estimated using the Kaplan-Meier estimator and 95% confidence intervals will be calculated using the logit transformation and the Greenwood variance estimate.
Overall survival (OS) | From initiation of treatment to death or last contact, whichever occurs first up to 2 years
  OS will be estimated using the Kaplan-Meier estimator and 95% confidence intervals will be calculated using the logit transformation and the Greenwood variance estimate.
PIPAC technical failure rate | Up to 2 years
  The technical failure rate will be calculated. The device malfunction rate will also be calculated. Rates and associated 95% Clopper and Pearson binomial confidence limits will be estimated.
Patient-reported health status and quality of life | At baseline and at 6, 12, 18 and 24 weeks off study
  Will be measured using the European Quality of Life Five Dimension Five Level Scale and will be summarized with descriptive statistics.
Patient-reported symptoms | At baseline and at 6, 12, 18 and 24 weeks off study
  Will be measured using the MD Anderson Symptom Inventory and will be summarized with descriptive statistics.
Time to peritoneal tumor associated complications | Up to 2 years
  Will be estimated using the Kaplan-Meier estimator and 95% confidence intervals will be calculated using the logit transformation and the Greenwood variance estimate.
Functional status | Up to 1 year
  Will be measured by the number of daily steps before and after treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Yanghee Woo, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States